CLINICAL TRIAL: NCT00570518
Title: DRUID Work Package 2 - Epidemiology
Brief Title: Alcohol and Other Psychoactive Substances in Road Traffic - a Case-control Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Collaborators: Hospital District of Helsinki and Uusimaa (Other); European Commission (Other)
Responsible Party: Sponsor
Other Study IDs: KTL 403-2; 404-3; 405-9; 406-5
Record Dates: First submitted 2007-12-10; First posted 2007-12-11 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-09

CONDITIONS: Prevalence of Psychoactive Substances in Road Traffic; Psychoactive Substances in Accident Involved Drivers; Relative Risk Estimation of Accident Involvement for Impaired Drivers
Keywords: driving under the influence; psychoactive substances; roadside surveys; hospital surveys; accident involvement risk estimation
MeSH Terms: conditions — Driving Under the Influence

STUDY DESIGN:
Observational Model: Case-Control
Biospecimen Retention: Samples With DNA — Whole blood and oral fluid are collected for the study. However, no DNA determinations are done at any point of the study. The laboratory where the samples are analysed does not analyse DNA. DNA is not relevant for this study.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: randomly stopped drivers of motorised vehicles and bicycles
- 2: drivers of motorised vehicles and bicycles injured or killed in road traffic accidents

SUMMARY:
The main purpose of the study is to determine the accident risk when driving under the influence of psychoactive substances, including alcohol (DUI). Other aims are to find out the prevalence of psychoactive substances in road traffic and to obtain information on the role of these substances in road traffic accident causations.

For the purposes of the study, drivers of motorised vehicles are randomly stopped and interviewed and breath alcohol is recorded. Also, an oral fluid sample is taken and psychoactive substances are investigated in the laboratory. For cases, drivers injured in traffic accidents are asked to participate to the study. A whole blood sample and, if possible, an oral fluid sample is taken and psychoactive substances are determined in the laboratory. Also, people diseased in road traffic accident are included in the study. The information required for these subjects are taken from a register database.

The study is part of an EU-project DRUID. Altogether 13 European countries take part to the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* driver of a motorised vehicle or bicycle
* is willing to participate to the study (not applicable to the diseased drivers; information obtained from a register database)

Exclusion Criteria:

* 17 or younger
* not the driver of a motorised vehicle or bicycle
* does not want to participate (not applicable to the diseased drivers; information obtained from a register database)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: drivers of motorised vehicles and bicycles in general road traffic or drivers of motorised vehicles and bicycles, injured or killed in road traffic accidents
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2007-09; Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
relative risk estimation of accident involvement for drivers impaired by psychoactive substances | three years

SECONDARY OUTCOMES:
prevalence of psychoactive substances in the general driving population | three years
prevalence of psychoactive substances among accident involved drivers | three years

CONTACTS AND LOCATIONS:
Overall Officials: Pirjo Lillsunde, Dr, Principal Investigator — National Public Health Institute
Locations (1):
- National Public Health Institute, Helsinki, Finland

REFERENCES:
- See also: The official homepage of the EU-project — http://www.druid-project.eu